CLINICAL TRIAL: NCT01880073
Title: Use of FemVue for Assessment of Tubal Patency as Compared to Laparoscopic Chromopertubation
Brief Title: FemVue and Tubal Patency
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1202012213
Record Dates: First submitted 2013-05-21; First posted 2013-06-18 (Estimated); Results first posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Tubal Patency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FemVue device (Experimental): FemVue would be used in conjunction with the laparoscopic chromopertubation to determine if it is as effective.
  Interventions: Device: FemVue device

INTERVENTIONS:
Device: FemVue device — The device will be used in conjunction with what is now considered the standard of care to determine if it's as effective.

SUMMARY:
A thorough infertility evaluation commonly involves determining whether a woman's fallopian tubes are patent. The two most often utilized methods of evaluating the fallopian tubes are hysterosalpingogram (taking an X-ray of the pelvis after injecting dye through the uterus and fallopian tubes) and laparoscopic chromopertubation (a surgical procedure in which dye is visualized passing through the fallopian tubes).

The FemVue Saline-Air device is a new method of assessing tubal patency. The device utilizes a mixture of saline and air bubbles that can be seen passing through the fallopian tubes by ultrasound. FemVue can be efficiently performed in a physician's office and is minimally invasive. Unlike hysterosalpingogram and laparoscopic chromopertubation, it does not carry the risks of anesthesia or surgery, and doesn't expose the patient to radiation or contrast. It does, like the other two methods, carry a small risk of infection.

This study will involve using the FemVue device on patients under anesthesia in the operating room before they undergo scheduled laparoscopic chromopertubation, the gold standard for evaluating tubal patency. The two methods will be compared to determine the accuracy of the FemVue device.

DETAILED DESCRIPTION:
Subjects who agree to participate will have their tubes evaluated by using the FemVue Saline-Air device and laparoscopic chromopertubation.

ELIGIBILITY:
Inclusion Criteria:

* Pts ages 18-45 undergoing planned diagnostic laparoscopy with chromopertubation.

Exclusion Criteria:

* Adnexal mass > 3.5cm or uterine size greater than 10 wks

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2016-05-24 (Actual); Study Completion 2019-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Spandorfer, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FemVue Device
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FemVue Device
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Had Concordant Findings
Description: When the findings using the device was the same as the procedure. In other words, if the device found tubes to be patent (open) and it was confirmed with the laparoscopic chromopertubation, the findings are said to be concordant the same as if the device found tubes to be blocked and the laparoscopic chromopertubation found the same.
Time Frame: End of procedure, day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | FemVue Device
Number analyzed (Participants) | 24
Participants | 21
Statistical Analysis 1: Comparison: FemVue Device; Test type: Other; Proportion = 0.875, 95% CI 2-sided [0.74 to 1.00]

2. Primary Outcome: Number of Subjects With Discordant Findings
Description: When the findings between the FemVue and Laparoscopic Chromopertubation were discordant, efficacy of FemVue was determined with a third procedure, a Hysterosalpingogram. If the FemVue device found the tubes patent (open) and laparoscopic chromopertubation found them closed, the finding is considered discordant. To determine which finding is accurate a third procedure was performed which is a Hysteropsalpingogram, another way to determine tubal patency.
Time Frame: End of procedure, day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | FemVue Device
Number analyzed (Participants) | 24
Participants | 3
Statistical Analysis 1: Comparison: FemVue Device; Test type: Other; Proportion = 0.125, 95% CI 2-sided [0.00 to 0.26]

3. Secondary Outcome: The Time Frame in Which Patency of the Tubes Was Determined With the FemVue Device.
Time Frame: 10 mins after start of procedure
Population: This information was not collected.
Arm/Group | FemVue Device
Number analyzed (Participants) | 0

4. Secondary Outcome: Time Frame in Which Patency of the Tubes Was Determined by Laparoscopic Chrompertubation.
Time Frame: End of procedure, Day 1
Population: This information was not collected.
Arm/Group | FemVue Device
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event was monitored for a 2 week period post procedure.
Arm/Group | FemVue Device
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

LIMITATIONS AND CAVEATS:
Limitations on study participants have precluded us from achieving statistically reliable results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No